CLINICAL TRIAL: NCT06232525
Title: A Randomized Comparison of Transobturator Tape With the Plication of Urethral Ligaments in the Treatment of Stress Urinary Incontinence
Acronym: added
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alev Esercan (Other Government)
Responsible Party: Sponsor-Investigator, Alev Esercan, Obstetrics and Gynecologist, MD, Sanliurfa Education and Research Hospital
Organization: Sanliurfa Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEAH-63
Record Dates: First submitted 2024-01-12; First posted 2024-01-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-01

CONDITIONS: Stress Incontinence, Female
Keywords: transobturator tape; urethral ligament plication
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: In the double-blind study, one group of patients with stress urinary incontinence will undergo transobturator tape surgery and the other group of patients will undergo urethral ligament plication surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients who are decided to have surgery due to stress urinary incontinence will undergo TOT surgery and urethral plication surgery, without being told which surgery they will have (both surgeries will be performed with the mid-urethral approach and the patient will not be told whether mesh is used or not), with a draw system in which the computer program will decide on the surgeon who will perform the surgery. The surgeon will always be the same person (Esercan A), and on the morning of the surgery, he will be told about the surgery he will perform and will be asked not to share it with the patient.
  At the end of the 5th day, 2.5 months, 6 months and 1 year after the surgery, patients will be called for a check-up and examined by the same doctor, different from the doctors who performed the surgery and wrote the publication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- transobturator tape operation group (Active Comparator): Patients who are decided to undergo surgery due to stress urinary incontinence are the group who will undergo TOT surgery through a lottery system where the computer program will decide on the surgeon who will perform the surgery, without being told which surgery they will have (both surgeries will be performed through the mid-urethral approach and the patient will not be told whether mesh is used or not).
  Interventions: Procedure: transobturator tape operation (TOT)
- urethral ligament plication group (Active Comparator): Patients who are decided to undergo surgery due to stress urinary incontinence are the group who will undergo urethral ligament plication surgery through a lottery system where the computer program will decide on the surgeon who will perform the surgery, without being told which surgery they will have (both surgeries will be performed through the mid-urethral approach and the patient will not be told whether mesh is used or not).
  Interventions: Procedure: urethral ligament plication

INTERVENTIONS:
Procedure: transobturator tape operation (TOT) — TOT surgery: With an 18 French Foley urinary catheter, the sling passes through the skin in the groin, the obturator foramen, the back of the adductor longus tendon, and the midurethral vaginal incision; extends 1 cm below the midpoint of the urethra, the tape is held in place without sutures by its interface with the patient's tissue. After the mesh is placed, the incision in the suburethral midline is closed.
  Arms: transobturator tape operation group
Procedure: urethral ligament plication — Urethral ligament plication: With an 18 French Foley urinary catheter, a vertical incision of approximately 3 cm is made in the anterior-lateral wall sulcus of the vagina on the right and left lines, 2 cm laterally from the midline, with the urethral meatus remaining in the midline, and external urethral ligaments on both sides inferolateral to the urethra, sutured in the midline by using 2-0 or 3-0 polyester sutures on both sides separately. The incised anterior vaginal tissue is closed one by one with 2-0 rapid Vicryl.
  Arms: urethral ligament plication group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of transobturator tape (TOT) operation and urethral ligament plication operation in stress incontinence patients. The main question:

* Which operation is more effective in treatment of stress incontinence?
* Which operation has less complication and risks? Participants will be followed about 5 days, 2.5 months, 6 months and 1 year after the operation and asked about the continence status and complications.

DETAILED DESCRIPTION:
The study will be a double-blind, prospective experimental study. When examining patients with stress urinary incontinence complaints, POP-Q staging in terms of pelvic organ prolapse before surgery, symptom interrogation in the examination of the anterior/middle and posterior compartments based on the Integral Theory in the pelvic floor examination, Urogenital Distress Inventory (UDI-6) for the evaluation of urinary incontinence and Female sexual function scale (FSFI) scales will be filled in to evaluate sexual functions. One group of patients will undergo transobturator tape (TOT), and the other group will undergo urethral ligament plication surgery.

Patients who are decided to have surgery due to stress urinary incontinence will undergo TOT surgery and urethral plication surgery, without being told which surgery they will have (both surgeries will be performed with the mid-urethral approach and the patient will not be told whether mesh is used or not), with a draw system in which the computer program will decide on the surgeon who will perform the surgery. The surgeon will always be the same person (Esercan A), and on the morning of the surgery, he will be told about the surgery he will perform and will be asked not to share it with the patient.

At the end of the 5th day, 2.5 months, 6 months and 1 year after the surgery, the patients were called for control and examined by the same doctor, different from the doctors who wrote the surgery and the publication. POP-Q staging was performed again in terms of pelvic organ prolapse, based on the Integral Theory in the pelvic floor examination. During the examination of the anterior/middle and posterior compartments, symptom inquiry, Urogenital Distress Inventory (UDI-6) for the evaluation of urinary incontinence and Female Sexual Function Scale (FSFI) scales will be filled in for the evaluation of sexual functions. The FSFI survey has 19 questions; It evaluates 6 main factors: sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain/discomfort. The highest total raw score that can be obtained in this scale is 95, the lowest raw score is 4, and after multiplying the coefficients, the highest score is 36 and the lowest score is 2. Impact coefficients used to score the entire scale; It was determined as 0.6 for sexual desire, 0.3 for sexual arousal and lubrication, and 0.4 for orgasm, satisfaction and pain/discomfort. A FSFI score below 26.55 is defined as compatible with sexual dysfunction. Additionally, if there are any complications, they will be recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years or older
2. Presence of stress urinary incontinence symptoms
3. Agreeing to have surgery

Exclusion Criteria:

1. Pregnancy
2. Being under 18 years of age
3. Suspicion of malignancy
4. History of previous mid-urethral sling or urinary incontinence surgery
5. Being diagnosed with intrinsic sphincter (urethral) insufficiency
6. Urinary incontinence due to neurological bladder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female urinary incontinence study
Enrollment: 108 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Subjective finding of no urinary incontinence | After the first day of the operation day and all of the follow-up (postoperative 5th day, 2.5 th month, 6th month and first year)
  The patient has no urinary incontinence and a significant decrease in the UDI-6 score.
Objective finding of no urinary incontinence | After the first day of the operation day and all of the follow-up(postoperative 5th day, 2.5 th month, 6th month and first year)
  Tap test negativity (if the patient's bladder is filled with 300cc physiological saline and the patient is made to cough and no urine leakage is observed, it is considered negative)

SECONDARY OUTCOMES:
complications | postoperative 5th day, 2.5 th month, 6th month and first year
  the presence of postoperative complications; Any complications such as presence of urinary incontinence, leg pain, inability to urinate, hematuria, pelvic organ injury

CONTACTS AND LOCATIONS:
Overall Officials: Peter Emanuel Petros, Prof., Study Director — retired; Alev Esercan, MD, Principal Investigator — Sanliurfa Education and Research Hospital
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)